CLINICAL TRIAL: NCT02401243
Title: A Pilot Descriptive Canadian, Multicenter, Open-label, Randomized Study of Two Titration Algorithms With Insulin Glargine 300 Units/mL in Type 2 Diabetes Mellitus Patients
Brief Title: Study of Two Titration Algorithms With Insulin Glargine 300 Units/mL in Type 2 Diabetes Mellitus Patients
Acronym: TITRATION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLARGL07496; U1111-1168-5158 (Other: UTN)
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (INSIGHT titration algorithm) (Experimental): INSULIN GLARGINE (U300): self-titration of insulin glargine 300 units/mL (U300) will be increased daily by 1 unit until fasting SMPG reaches the target range of 4.4 to 5.6 mmol/L
  Interventions: Drug: INSULIN GLARGINE (U300)
- Cohort 2 (EDITION titration algorithm) (Experimental): INSULIN GLARGINE (U300): titration of insulin glargine 300 units/mL (U300) will be adjusted weekly or not more than every 3 days to achieve the target range of fasting SMPG of 4.4 to 5.6 mmol/L
  Interventions: Drug: INSULIN GLARGINE (U300)

INTERVENTIONS:
Drug: INSULIN GLARGINE (U300) — Pharmaceutical form: pre-filled disposable pen
  Route of administration: subcutaneous
  Other Names: HOE901

SUMMARY:
Primary Objective:

The primary objective of this study is to obtain efficacy and safety descriptive data on 2 different titration algorithms: the INSIGHT titration algorithm (self-titration of 1 unit/day) and the EDITION trial algorithm with insulin glargine 300 units/mL when given as basal insulin in uncontrolled type 2 diabetes mellitus (T2DM) patients on basal insulin with or without non-insulin anti-hyperglycemic agent (NIAHA) or in insulin naïve patients.

Secondary Objective:

The secondary objective is to gain additional efficacy and safety data (glycated hemoglobin [A1C], fasting plasma glucose [FPG], 7-point self-measure plasma glucose [SMPG], insulin dose and weight) and determine patient related outcome and health care professional satisfaction as it pertains to each titration regimen.

DETAILED DESCRIPTION:
The total study duration is approximately 14 weeks (2 weeks screening and 12 weeks treatment) with a 2-day safety follow-up and a study extension of 12 weeks for eligible patients.

ELIGIBILITY:
Inclusion criteria:

* Patients with type 2 diabetes mellitus.
* Patients who are ≥18 years of age.
* Treated for diabetes for at least 6 months.

  * If on basal insulin, stable for at least 3 months prior to screening visit on their basal insulin treatment(s) (±20% total insulin dose)
  * If on NIAHA, stable for at least 8 weeks prior to screening visit on their NIAHA(s) (no change in dose or initiation of new NIAHAs).
* Patients on uncontrolled basal insulin (insulin glargine, normal protamine Hagedorn [NPH], detemir) +/ NIAHAs with an A1c >7.0% and ≤10% or uncontrolled on NIAHAs (insulin naïve patients) with an A1c >7.0% and ≤11%.
* Signed informed consent form.

Exclusion criteria:

* Patients with type 1 diabetes mellitus (T1DM).
* Nightshift worker.
* Female patients who are pregnant or lactating.
* Treatment with an insulin other than basal insulin (premixes, rapid insulin, fast acting insulin analogues) within the previous 3 months.
* Patients with less than 1 year history of diabetes.
* Patients unwilling to inject insulin or perform self-monitoring blood glucose.
* Current alcohol or drug abuse.
* Patients unlikely to comply with the protocol and complete the study eg, uncooperative attitude, inability to return for follow-up visits.
* Patients with active cancer or any other diseases or conditions which in the opinion of the Investigator would make the patient unsuitable for participation in the study.
* Any clinically significant laboratory findings that in the judgment of the Investigator would preclude safe completion of the study.
* Known allergies to study drugs.
* Participation in another clinical study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching fasting SMPG ≤5.6 mmol/L without nocturnal (midnight to 6:00 am) hypoglycemia (confirmed or symptomatic or severe) | 12 weeks

SECONDARY OUTCOMES:
Percentage of patients with adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (25):
- Canada (25):
  - Investigational Site Number 124001, Abbotsford
  - Investigational Site Number 124013, Brampton
  - Investigational Site Number 124008, Burlington
  - Investigational Site Number 124024, Burnaby
  - Investigational Site Number 124015, Collingwood
  - Investigational Site Number 124025, Corunna
  - Investigational Site Number 124019, Etobicoke
  - Investigational Site Number 124021, Hamilton
  - Investigational Site Number 124011, Laval
  - Investigational Site Number 124005, Lévis
  - Investigational Site Number 124018, London
  - Investigational Site Number 124003, Oshawa
  - Investigational Site Number 124010, Québec
  - Investigational Site Number 124012, Québec
  - Investigational Site Number 124007, Sarnia
  - Investigational Site Number 124002, Saskatoon
  - Investigational Site Number 124023, Sherbrooke
  - Investigational Site Number 124009, Smiths Falls
  - Investigational Site Number 124017, Strathroy
  - Investigational Site Number 124020, Toronto
  - Investigational Site Number 124006, Vancouver
  - Investigational Site Number 124026, Vancouver
  - Investigational Site Number 124004, Victoria
  - Investigational Site Number 124014, Winnipeg
  - Investigational Site Number 124016, Winnipeg